CLINICAL TRIAL: NCT01952041
Title: A New Paradigm for Illness Monitoring and Relapse Prevention in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH103148-01 D14022
Record Dates: First submitted 2013-09-20; First posted 2013-09-27 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Mobile Application; Relapse; SMI; EHealth; E-Health; Health Technology; mHealth; m-Health; Mobile Health; Serious Mental Illness; Electronic Health
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Recurrence | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded clinical assessors also conducted assessments with all participants at baseline and every 3 months post-randomization.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device: Smartphone (Experimental): Participants in the smartphone intervention arm received treatment as usual in addition to receiving a smartphone with the study application. The study application identified relapse risk and prompted the clinical team to provide enhanced services.
  Interventions: Behavioral: Device: Smartphone
- Treatment as Usual (Active Comparator): Treatment as usual included outpatient case management, linkage to services and medication monitoring.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Device: Smartphone
  Arms: Device: Smartphone
Behavioral: Treatment as usual
  Arms: Treatment as Usual

SUMMARY:
This study was a 2-arm randomized control trial (RCT) designed to test a multi-modal smartphone data collection system that provided mobile monitoring of schizophrenia to detect early signs of relapse. The RCT compared an arm with participants who received treatment as usual with an arm that received the smartphone system for a year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) criteria for schizophrenia, schizoaffective disorder, or psychosis not otherwise specified based on a chart diagnosis
* 18 years or older
* An inpatient psychiatric hospitalization, daytime psychiatric hospitalization, outpatient crisis management, or short-term psychiatric hospital emergency room within 12 months before study entry
* Willing and able to provide informed consent

Exclusion Criteria:

* Hearing, vision, or motor impairment that make it impossible to operate a smartphone (determined using a demonstration smartphone for screening)
* 6th grade reading level (determined by Wide Range Achievement Test- 4th Edition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2015-03-13 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dror Ben-Zeev, PhD, Principal Investigator — University of Washington
Locations (1):
- Zucker Hillside Hospital, Glen Oaks, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible individuals at a medical clinic were identified through electronic medical records and approached by a staff member to be recruited for the study. Recruitment was open from March 2015 until July 2016.
Pre-assignment Details: N=23 participants withdrew before randomization:
  N=1 did not complete baseline, N=15 no longer receiving services at the study site, N=1 incarcerated, N=6 no longer interested in participating.
Period: Overall Study
Arm/Group | Device: Smartphone | Treatment as Usual
Started | 62 | 64
Completed | 45 | 43
Not Completed | 17 | 21
Not completed — Lost to Follow-up | 9 | 16
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Device: Smartphone | Treatment as Usual | Total
Number analyzed (Participants) | 62 | 64 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (14) | 36 (13) | 37 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 54
  Male | 36 | 36 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 15 | 32
  Not Hispanic or Latino | 45 | 49 | 94
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 8 | 9
  Native Hawaiian or Other Pacific Islander | 4 | 2 | 6
  Black or African American | 18 | 16 | 34
  White | 23 | 21 | 44
  More than one race | 13 | 15 | 28
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Relapses in Participants
Description: A count of participants who experienced relapse, as defined as one of the following events: psychiatric hospitalization, a significant increase in the level of psychiatric care (i.e. frequency and intensity of services), an increase in medication in addition to a 25% increase in Brief Psychiatric Rating Scale (BPRS) from last assessment, suicidal or homicidal ideation that was clinically significant in the investigator's judgement, deliberate self-injury, violent behavior resulting in damage to another person or property.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Smartphone | Treatment as Usual
Number analyzed (Participants) | 62 | 64
Participants | 20 | 22
Statistical Analysis 1: Comparison: Device: Smartphone vs Treatment as Usual; Test type: Superiority; p = 0.80, Chi-squared; Chi-square test statistic=0.06, degrees of freedom=2

2. Primary Outcome: Time to Relapse
Description: Time to first relapse was defined as the time from randomization until the first relapse. Participants who did not experience a relapse were censored at their last known time relapse-free. Time-to-first relapse was estimated using the Kaplan-Meier method.
Time Frame: From randomization date until first relapse (evaluated approximately every 3 months until their last study visit which occurred approximately 12 months from randomization for those who completed the study).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Device: Smartphone | Treatment as Usual
Number analyzed (Participants) | 62 | 64
months | 13.8 [NA to NA] — Not enough participants relapsed to calculate the upper and lower 95% confidence interval (CI). | NA [9.7 to NA] — In the treatment as usual group (TAU), the median from the time-to-event analysis was not reached (that is, at least 50% of people did not relapse). Not enough participants relapsed to calculate the upper 95% confidence interval (CI).
Statistical Analysis 1: Comparison: Device: Smartphone vs Treatment as Usual; Test type: Superiority; p = 0.43, Regression, Cox; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.42 to 1.44] — Hazard ratio is intervention arm vs. TAU for time to first relapse from randomization. There is not a standard error (SE) that directly links to the hazard ratio. The confidence interval provided illustrates the dispersion for the hazard ratio

3. Secondary Outcome: Psychotic Symptom Severity
Description: Psychotic symptom severity assessed using the Brief Psychiatric Rating Scale (BPRS). This is an 18-item scale that rates severity of positive symptoms (including auditory hallucinations and persecutory ideation), and mood and behavioral symptoms. Items are rated by a clinical assessor on a scale of 1 (absent) to 7 (very severe). Total scores range from 18-126. Higher scores indicate worse symptoms.
Time Frame: Assessed at baseline and every three months for one year.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Device: Smartphone | Treatment as Usual
Number analyzed (Participants) | 62 | 64
score on a scale
  baseline | 26.3 (7.2) | 27.4 (8.2)
  3 months | 24.9 (6.4) | 25.3 (5.3)
  6 months | 25.3 (6.5) | 23.7 (5.1)
  9 months | 25.6 (6.4) | 24.0 (5.6)
  12 months | 25.0 (7.7) | 26.3 (8.5)
Statistical Analysis 1: Comparison: Device: Smartphone vs Treatment as Usual; Test type: Superiority; p = 0.58, Mixed Models Analysis; Slope = 0.22, 95% CI 2-sided [-0.58 to 1.02], Standard Error of Mean 0.41 — Treatment by time interaction terms are given to test difference of slopes between arms

4. Secondary Outcome: Depression
Description: Depression measured using the Calgary Depression Scales (CDSS). This is a 9-item assessment with values of 0 (absent) to 3 (severe) of depressive symptoms separate from positive, negative and extrapyramidal symptoms in people with schizophrenia. Total scores range from 0-27. A higher score indicates more severe symptoms.
Time Frame: Assessed at baseline and every three months for one year.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Device: Smartphone | Treatment as Usual
Number analyzed (Participants) | 62 | 64
score on a scale
  baseline | 1.4 (2.0) | 2.1 (2.7)
  3 months | 1.7 (2.2) | 1.7 (2.1)
  6 months | 1.4 (2.3) | 1.7 (2.3)
  9 months | 2.1 (2.6) | 1.7 (2.0)
  12 months | 1.4 (2.2) | 2.5 (2.5)
Statistical Analysis 1: Comparison: Device: Smartphone vs Treatment as Usual; Test type: Superiority; p = 0.84, Mixed Models Analysis; Slope = 0.02, 95% CI 2-sided [-0.22 to 0.26], Standard Error of Mean 0.12 — Treatment by time interaction terms are given to test difference of slopes between arms

5. Secondary Outcome: Social Functioning
Description: Social Functioning was assessed using the Social Functioning Scale (SFS). This is a 76-item questionnaire that assesses various aspects of social functioning and generates a number of subscale scores including social withdrawal, interpersonal behavior, pro-social activities, and an overall score of social functioning. The item values range from 0 (almost never) to 3 (often). Total scores range from 0-228. A higher score indicates greater social functioning.
Time Frame: Assessed at baseline and every three months for one year.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Device: Smartphone | Treatment as Usual
Number analyzed (Participants) | 62 | 64
score on a scale
  baseline | 142.0 (29.0) | 135.1 (30.2)
  3 months | 144.9 (30.3) | 140.0 (27.2)
  6 months | 145.8 (27.2) | 140.1 (28.1)
  9 months | 134.5 (30.5) | 143.2 (28.0)
  12 months | 138.1 (27.9) | 141.1 (26.1)
Statistical Analysis 1: Comparison: Device: Smartphone vs Treatment as Usual; Test type: Superiority; p = 0.06, Mixed Models Analysis; Slope = -2.70, 95% CI 2-sided [-5.40 to 0.04], Standard Error of Mean 1.40 — Treatment by time interaction terms are given to test difference of slopes between arms

ADVERSE EVENTS:
Time Frame: Data was collected for each participant at baseline and every 3 months for 1 year.
Arm/Group | Device: Smartphone | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 1/62 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/64
Other Adverse Events (participants affected / at risk) | 0/62 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT01952041/Prot_SAP_000.pdf